CLINICAL TRIAL: NCT03180593
Title: A Prospective, Randomized, Open-Label, 13 to 14-week Study of the Efficacy and Safety of Valsartan and Nebivolol/Valsartan in Hypertensive Subjects With Left Ventricular Hypertrophy (LVH)
Brief Title: Efficacy and Safety of Valsartan and Nebivolol/Valsartan in Hypertensive Patients With LVH
Acronym: BVreduce
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Trinity Hypertension & Metabolic Research Institute (Other)
Collaborators: Allergan Sales, LLC (Industry)
Responsible Party: Principal Investigator, Henry Anthony Punzi, Director of Clinical Research, Trinity Hypertension & Metabolic Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BYS-IT-78
Record Dates: First submitted 2017-06-06; First posted 2017-06-08 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Hypertension Complicated; Hypertrophy, Left Ventricular; Blood Pressure
MeSH Terms: conditions — Hypertrophy, Left Ventricular | interventions — Valsartan; Nebivolol

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, open label, blinded-endpoint (PROBE)
Who Masked: Investigator
Masking Description: alternating
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Valsartan Arm (Active Comparator): Valsartan 80mg randomly assigned for 8 weeks to asses BP control with office and 24-hour ABPM and reduction of LVH
  Interventions: Drug: Valsartan 80 mg
- Nebivolol/Valsartan (Active Comparator): Nebivolol/Valsartan 5/80mg randomly assigned for 8 weeks to asses Blood Pressure control with office and 24-hour Ambulatory Blood Pressure Monitoring and reduction of Left Ventricular Hypertrophy
  Interventions: Drug: Valsartan 80 mg

INTERVENTIONS:
Drug: Valsartan 80 mg — Compare office and 24-hour Blood Pressure Control and regression of Left Ventricular Hypertrophy
  Other Names: Nebivolol/Valsartan 5/80mg

SUMMARY:
To assess the efficacy of Left Ventricular Hypertrophy (LVH) reduction and 24-hour blood pressure control of Valsartan 80mg or Nebivolol/Valsartan 5/80mg once daily as replacement therapy for currently treated or untreated hypertensive patients with LVH not at BP goal.

DETAILED DESCRIPTION:
The potential benefits of blood pressure reduction have been demonstrated in numerous large clinical trials. The most recent is the SPRINT Trial demonstrating that lower blood pressure goals can be achieved and are associated with a significant decrease in morbidity and mortality. The latest NHANES 2012 data reveal that less than 50% of patients that are aware of the elevated blood pressure and are being treated achieve blood pressure control. Treatment of hypertension in many patients (>70%) require treatment with more than one drug, increasing the likelihood of non-compliance and not achieving blood pressure goal. JNC 8 recommends the utilizing of combination therapy both for Stage I and Stage II Hypertensive patients.

Objectives of the study to assess the efficacy of LVH reduction and 24-hour blood pressure control of Valsartan 80mg and Nebivolol/Valsartan 5/80mg, once daily for the treatment of currently treated hypertensive patients with LVH.

The study will evaluate LVH reduction at 4 and 8 weeks as well as change from baseline in mean 24 hour ABPM SBP after 4 and 8 weeks of treatment with valsartan 80mg or nebivolol/valsartan 5/80mg

ELIGIBILITY:
Inclusion Criteria:

1. Capable of reading, comprehending the consent process and providing written informed consent to participate in the study.
2. Male or female ≥ 18 years of age who are either newly diagnosed with HTN or who are currently being treated.
3. Patients must have a mean cuff sitting diastolic blood pressure cuff (DBP) > 90 mmHg and <105 mmHg (< 100 mmHg on prior treatment) and mean cuff sitting systolic blood pressure (SBP) <160 mmHg, at two consecutive qualifying visits during the placebo run in period.
4. Arm circumference < 45cm.
5. Compliance with single blind placebo capsules between V1 to 4 or 4X of 80-120%.
6. Women may be enrolled if the following criteria are met:

1.- Have a negative serum pregnancy test at screening 2.- Are not breastfeeding 3.- Do not plan to become pregnant during the study 4.- Have had a hysterectomy or tubal ligation at least 6 months prior to signing the informed consent form or 5.- Have been postmenopausal for at least 1 year or 6. - If they are of childbearing potential and will practice one of the following methods of birth control throughout the study: oral, patch, injectable, or implantable hormone contraception, intrauterine device, diaphragm plus spermicide or female condom plus spermicide. Abstinence, partner's vasectomy are not acceptable methods of contraception.

7. Diagnosis of Left Ventricular Hypertrophy (LVH).

Exclusion Criteria:

1. Known allergy or hypersensitivity to Beta-Blockers.
2. Known allergy or hypersensitivity to Angiotensin II Receptor Blockers.
3. Patients with severe hypertension (mean seated cuff DBP>115 mmHg or mean seated SBP> 180mmHg) or any form of secondary hypertension.
4. Patients within the past 6 months with a history of hypertensive encephalopathy, stroke or transient ischemic attack.
5. Patients within the last 6 months with a history of myocardial infarction, percutaneous transluminal coronary revascularization, coronary bypass graft, valvular surgery or unstable angina.
6. Patients with evidence of resting bradycardia (<50 bpm) via palpation.
7. Patients with a history of heart block greater than First Degree Sino-atrial Block. Wolff-Parkinson-White Syndrome, Sick Sinus Syndrome, Atrial Fibrillation, Atrial Flutter, Congestive Heart Failure, or other manifestations of clinically significant cardiac valvular disease.
8. Patients with hemodynamically significant cardiac valvular disease.
9. Patients with evidence of significant chronic renal impairment as indicated by a serum creatinine of > 2.5mg/dL.
10. Patients with evidence of liver disease as indicated by AST (SGOT) or ALT (SGPT) > 2.5 times or total bilirubin > 1.5 times, the upper limit of the laboratory normal range.
11. Patients who demonstrate other laboratory test values deviating from the normal range which are considered to be clinically significant by the investigator.
12. Patient with a history or presence of gastrointestinal disease which may interfere with drug absorption.
13. Patients with insulin and non-insulin dependent diabetes mellitus not controlled on diet, insulin, or oral hypoglycemics as defined by a HgA1c >10.
14. Severe psychological or emotional condition which may interfere with participation in the study.
15. History of or current use of illicit drugs or alcohol abuse.
16. Participation in a clinical trial and taking any investigational drug within 30 days prior to enrolling into the study (Screening Visit).
17. A physical condition that would limit accurate BP measurement.
18. Inability to swallow a tablet or capsule.
19. History of moderate or severe asthma or COPD.
20. Any other medical condition which, in the Investigator's opinion, may render the patient unable to complete the study or which would interfere with optimal participation in the study or produce significant risk to the patient.
21. Patients taking more than two blood pressure medications
22. Patients currently taking a beta blocker

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2018-01-25 (Actual); Study Completion 2018-01-25 (Actual)

PRIMARY OUTCOMES:
LVH reduction at 4 weeks. | 4 weeks
  Reduction of Left ventricular hypertrophy from baseline compared to 4 weeks of treatment
24hr-ABPM measurement Change from baseline in mean 24 hour ABPM SBP | 4 weeks
  Reduction of Systolic BP over 24 hours baseline compared to 4 weeks of treatment

SECONDARY OUTCOMES:
LVH reduction at 8 weeks. | 8 weeks
  Reduction of Left ventricular hypertrophy from baseline compared to 8 weeks of treatment
24hr-Systolic ABPM measurement | 8 weeks
  Reduction of Systolic BP over 24 hours baseline compared to 8 weeks of treatment
24hr- DBP ABPM measurements | 4 and 8 weeks
  Mean change from baseline in trough DBP after 4 and 8 weeks of treatment with valsartan 80mg or nebivolol/valsartan 5/80mg
Office Blood Pressure measurements | 4 and 8 weeks
  Mean change from baseline in trough SBP after 4 and 8 weeks of treatment with valsartan 80mg or nebivolol/valsartan 5/80mg

CONTACTS AND LOCATIONS:
Overall Officials: Henry A Punzi, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Trinity Hypertension & Metabolic Research Institute, Carrollton, Texas, United States

IPD SHARING:
Plan to Share IPD: No